CLINICAL TRIAL: NCT00461890
Title: Long-Acting Injectable Naltrexone Treatment of Alcohol Dependence in Primary Care vs. in Specialized Chemical Dependence Treatment: A Pilot Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Batki, M.D., Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Syracuse VA IRB #00364
Record Dates: First submitted 2007-04-13; First posted 2007-04-18 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Alcohol Dependence; Veterans
Keywords: Alcohol; Veterans; Primary Care; Naltrexone
MeSH Terms: conditions — Alcoholism

INTERVENTIONS:
Drug: Injectable Naltrexone

SUMMARY:
The goal of the proposed project is to improve the primary care treatment of veterans with alcohol dependence. Alcohol dependence is a common behavioral health problem among veterans treated in VA primary care clinics. However, assessment and treatment of alcohol dependence in primary care remains problematic. Assessment of veterans with positive alcohol use screens may not always be completed and referrals to specialty care may not always be made. Moreover, the use of medications for alcohol dependence among veterans is rare, despite VA treatment guidelines that recommend such use. Finally, when medications are prescribed, patients may have difficulties with adherence.

The primary aim of this study is to assess the feasibility of long-acting injectable naltrexone provided through primary care (LAN/PC) versus long-acting injectable naltrexone in the specialized chemical dependence clinic (LAN/CDC). The secondary aim is to obtain preliminary assessments of the relative effectiveness of long-acting injectable naltrexone in primary care versus in the chemical dependence clinic.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or non-pregnant females between the ages of 18 and 69 who are receiving their primary medical care at the Syracuse VAMC.
* Participants must meet DSM-IV diagnostic criteria for current alcohol dependence.
* Participants must report drinking within the thirty days prior to study entry.
* Participants must receive approval from their primary care provider for study participation.
* Participants must be willing to consider accepting at least one of the two treatment conditions.

Exclusion Criteria:

* Participants with a current DSM-IV diagnosis of current opioid abuse or dependence, or in opioid withdrawal
* AST level is greater than 3 times the upper limit of the normal range
* Participants with a medical condition requiring opioid medication or a severe allergy to naltrexone
* Participants who received outpatient treatment at the Syracuse VA Chemical Dependence Clinic in the past 90 days
* Any unstable medical or psychiatric conditions in the judgment of the principal investigator or the participants primary care provider

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: Feasibility of an injectable naltrexone study in the primary care setting.

SECONDARY OUTCOMES:
Secondary Outcome: Effectiveness of long-acting injectable naltrexone in primary care versus in the chemical dependence clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Batki, M.D., Principal Investigator — Executive Director VA Center for Integrated Healthcare, Syracuse VA Medical Center
Locations (1):
- Syracuse VAMC, Syracuse, New York, United States